CLINICAL TRIAL: NCT05253456
Title: Modified Tubularized Incised Plate Urethroplasty (Snodgrass) For Distal Hypospadias Repair in a Circumcised Patient With the Use of a Derma -Dartos Flap for Second Layer Closure: Our Initial Experience
Brief Title: Modified Second Layer Repair for Distal Penile Hypospadias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, Assistant lecturer, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R22/2018
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): patients underwent our newly modified technique for hypospadias repair
  Interventions: Procedure: Derma -Dartos Flap for second layer closure

INTERVENTIONS:
Procedure: Derma -Dartos Flap for second layer closure — usage of Derma -Dartos Flap for second layer closure of a distal penile hypospadias in circumcised patients

SUMMARY:
to evaluate a modification to snodgrass technique in second layer closure of distal penile hypospadias

DETAILED DESCRIPTION:
In our study, we applied a new modification by using an intervening layer of a de-epithelialized ventral derma-dartos flap for neourethral covering. we present our newly applied technique and its impact on the success rate.

ELIGIBILITY:
Inclusion Criteria:

* All male patient with distal penile hypospadias aged less than 18

Exclusion Criteria:

* Patients with penile rotation or hypoplastic urethral plate were excluded from the study

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Hypospadias is congenital urethra defect in male urethra only
Enrollment: 102 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
urethro-cutaneous fistula | 1 year follow up
  presence of urethro-cutaneous fistula after closure of hypospadias as assess by inspection for the presence of urinary fistula

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No